CLINICAL TRIAL: NCT00953888
Title: A Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral AZD5069 After Single Ascending Doses in Healthy Male and/or Female Subjects
Brief Title: Study to Investigate the Safety, Tolerability and Activity of AZD5069 When Given as a Single Dose to Healthy Male and/or Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D3550C00001
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
Keywords: Healthy volunteer; Single ascending dose; Safety; Tolerability; Healthy volunteer study
MeSH Terms: interventions — N-(2-(2,3-difluoro-6-benzylthio)-6-(3,4-dihydroxybutan-2-yloxy)pyrimidin-4-yl)azetidine-1-sulfonamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Active (Experimental): AZD5069 oral solution
  Interventions: Drug: AZD5069
- Placebo (Placebo Comparator): Placebo oral solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD5069 — Single dose of oral solution.
  Arms: Active
Drug: Placebo — Single dose of oral solution.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine how well tolerated and safe AZD5069 is at different dose levels in healthy male and/or females. The study will also investigate how quickly AZD5069 is absorbed into and cleared by the body.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent
* Healthy male or female (of non child bearing potential) caucasian subjects aged 18 to 65 years with suitable veins for cannulation or repeated venepuncture
* Body mass index of between 18 and 30 kg/m2 inclusive

Exclusion Criteria:

* Subjects must not have any clinically significant disease or disorder, which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results, or the subjects ability to participate in the study
* Subjects must not have any history of gastrointestinal, liver or kidney disease, or any other condition known to interfere with how drugs are absorbed, used or eliminated by the body
* Subjects must not have had any significant illness or medical/surgical procedures or injuries with 4 weeks of administration of the investigational product

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of AZD5069 assessing vitals signs (blood pressure, pulse rate,body temperature), ECG,laboratory variables (including high sensitivity C-reactive protein, circulating neutrophils), continuous cardiac monitoring using telemetry. | Baselines assessments at Visit 1 (enrolment). Assessments pre-dose at Visit 2 and at protocol defined time-points post-dose. Follow up assessments at Visit 3.

SECONDARY OUTCOMES:
Pharmacokinetic profile: concentration of AZD5069 in blood | Samples collected at Visit 2 from pre-dose and at regular protocol defined intervals up to 96 hours post-dose.
Measurement of the effect of AZD5069 on circulating neutrophils | Samples collected at Visit 2 from pre-dose and at regular protocol defined intervals up to 96 hours post-dose.
Pharmacodynamic profile: assessment of ex vivo GROa stimulated CD11b expression on neutrophils in whole blood | Samples collected at Visit 2 from pre-dose and at regular protocol defined intervals up to 48 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sparrow, BSc, BMedSci, BM,BS, Principal Investigator — AstraZeneca Clinical Pharmacology Unit, Queens Medical Centre, Nottingham NG7 2UH
Locations (1):
- Research Site, Nottingham, United Kingdom

REFERENCES:
- [Derived] Cullberg M, Arfvidsson C, Larsson B, Malmgren A, Mitchell P, Wahlby Hamren U, Wray H. Pharmacokinetics of the Oral Selective CXCR2 Antagonist AZD5069: A Summary of Eight Phase I Studies in Healthy Volunteers. Drugs R D. 2018 Jun;18(2):149-159. doi: 10.1007/s40268-018-0236-x. PMID 29856004
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1335&filename=D3550C00001_Study_Synopsis.pdf